CLINICAL TRIAL: NCT00073437
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial Evaluating the Safety and Efficacy of Infliximab (Remicade�) in Subjects With Chronic Sarcoidosis With Pulmonary Involvement.
Brief Title: A Study of Infliximab in Patients With Sarcoidosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005293
Record Dates: First submitted 2003-11-20; First posted 2003-11-24 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Sarcoidosis
Keywords: Sarcoidosis; Infliximab; Pulmonary involvement; Remicade
MeSH Terms: conditions — Sarcoidosis | interventions — Infliximab

INTERVENTIONS:
Drug: Infliximab

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of infliximab (Remicade) in patients with Chronic Sarcoidosis. Infliximab (Remicade) targets specific proteins in the body's immune system to help control the development of inflammation to help reduce painful disease.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and effectiveness of infliximab in the treatment of subjects with sarcoidosis with pulmonary involvement who show symptoms of the disease even though they are currently being treated with medication. Patients will receive either placebo, 3 mg/kg infliximab, or 5 mg/kg infliximab infusions at weeks 0, 2, 6, 12, 18, and 24. Safety evaluations will be performed at specified intervals throughout the study and will consist of laboratory tests, vital signs (such as blood pressure), physical examinations and the occurrence and severity of adverse events as well as other study specific procedures. Patients will receive infusions of Infliximab (Remicade) 3 or 5 mg/kg or placebo at weeks 0, 2, 6, 12, 18 and 24.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been diagnosed with sarcoidosis at least 1 year prior to entry into the study
* Patients must have laboratory test diagnosing sarcoidosis prior to screening
* Patients must have a diagnosis of sarcoidosis by chest x- ray

Exclusion Criteria:

* Patients must not have used any investigational drug within 1 month prior to entering the study
* Patients must not have received previous administration of a treatment with any other therapeutic agent targeted at reducing TNF such as pentoxifylline, thalidomide, etanercept, CDP 870, adalimumab, within 3 months prior to screening
* Patients must not have received vaccinations within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2003-10; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the percent of predicted Full Vital Capacity (FVC) at week 24

SECONDARY OUTCOMES:
Change from baseline in Saint George's Respiratory Questionnaire total score, Change from baseline in the 6-minute walk distance, Change from baseline in Borg's CR10 dyspnea score, proportion of LuPGA responders at week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Baughman RP, Drent M, Kavuru M, Judson MA, Costabel U, du Bois R, Albera C, Brutsche M, Davis G, Donohue JF, Muller-Quernheim J, Schlenker-Herceg R, Flavin S, Lo KH, Oemar B, Barnathan ES; Sarcoidosis Investigators. Infliximab therapy in patients with chronic sarcoidosis and pulmonary involvement. Am J Respir Crit Care Med. 2006 Oct 1;174(7):795-802. doi: 10.1164/rccm.200603-402OC. Epub 2006 Jul 13. PMID 16840744
- [Result] Judson MA, Baughman RP, Costabel U, Flavin S, Lo KH, Kavuru MS, Drent M; Centocor T48 Sarcoidosis Investigators. Efficacy of infliximab in extrapulmonary sarcoidosis: results from a randomised trial. Eur Respir J. 2008 Jun;31(6):1189-96. doi: 10.1183/09031936.00051907. Epub 2008 Feb 6. PMID 18256069
- [Derived] Sweiss NJ, Barnathan ES, Lo K, Judson MA, Baughman R; T48 Investigators. C-reactive protein predicts response to infliximab in patients with chronic sarcoidosis. Sarcoidosis Vasc Diffuse Lung Dis. 2010 Jul;27(1):49-56. PMID 21086905
- [Derived] Baughman RP, Shipley R, Desai S, Drent M, Judson MA, Costabel U, du Bois RM, Kavuru M, Schlenker-Herceg R, Flavin S, Lo KH, Barnathan ES; Sarcoidosis Investigators. Changes in chest roentgenogram of sarcoidosis patients during a clinical trial of infliximab therapy: comparison of different methods of evaluation. Chest. 2009 Aug;136(2):526-535. doi: 10.1378/chest.08-1876. Epub 2009 Apr 24. PMID 19395578
- See also: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial Evaluating the Safety and Efficacy of Infliximab (REMICADE�) in Subjects with Chronic Sarcoidosis with Pulmonary Involvement — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=161&filename=CR005293_CSR.pdf